CLINICAL TRIAL: NCT02135211
Title: Feasibility and Acceptability of a Lifestyle Intervention for Patients Receiving Surgical Treatment for Lung Surgery
Brief Title: Healthy Directions After Lung Surgery Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Mary E. Cooley, Phd, Nurse Scientist, PhD, CRNP, FAAN, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-150
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: non-small cell lung cancer (NSCLC); multiple risk factor; lifestyle intervention; health behavior; lifestyle risk reduction; health related quality of life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Health Behavior; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): This is a single arm, quasi-experimental, pre- and post- test study design to test the feasibility and acceptability of a multiple risk factor, lifestyle intervention in patients receiving surgical treatment for lung cancer or those suspected of having lung cancer.
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling

SUMMARY:
The objective of this proposal is to test the feasibility and acceptability of a lifestyle risk reduction intervention for patients with lung cancer receiving surgical treatment. This study will provide the preliminary data needed to conduct a larger randomized controlled trial that tests an innovative, multidisciplinary intervention that has the potential to transform the standard of care for patients receiving surgical treatment for lung cancer.

ELIGIBILITY:
Patient Inclusion Criteria:

* > 21 years of age
* English speaking
* MD approval to participate in study
* Meets one of the inclusions below:
* 1. a histological diagnosis of NSCLC undergoing potentially curative treatment
* 2. OR those undergoing surgical procedures for lung cancer (includes patients undergoing diagnostic testing or those presenting with lung nodules
* 3.OR patients who have had a surgical procedure for lung cancer within the last six months.
* May invite a buddy to join study with them defined as a friend, partner, adult child or sibling

Buddy Inclusion Criteria:

* ≥ 21 years of age,
* English speaking, who is invited by the subject to join as a support person (e.g., friend, partner, adult child or sibling)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability | at end of study (4 months post intervention)
  The primary outcome measures to establish feasibility and acceptability of the intervention for this study are enrollment rates.
Feasibility and acceptability | at end of study (4 months post intervention)
  The primary outcome measures to establish feasibility and acceptability patient's use of intervention materials
Feasibility and acceptability | at end of study (4 months post intervention
  The primary outcome measures to establish feasibility and acceptability of the completion of self-monitoring
Feasibility and acceptability | at end of study (4 months post intervention)
  The primary outcome measures to establish feasibility and acceptability of the intervention for this study completion of nurse-patient contacts.

SECONDARY OUTCOMES:
Interest for this study | baseline, 1 month, & 4 month
  The secondary outcome measures of interest for this study are lifestyle risk reduction and Health Related-Quality of Life.
Interest for this study | baseline, 1 month, & 4 month
  The secondary outcome measures of interest for this study is an interview to evaluate the intervention will be conducted with the participant and the partner at the conclusion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Cooley, PhD, RN, FAAN, Principal Investigator — Dana Farber Cancer Insitute
Locations (2):
- United States (2):
  - Brigham & Woman's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts